CLINICAL TRIAL: NCT00873587
Title: Randomized Clinical Trial Evaluating the Optimal Technique for Chest Tube Removal
Brief Title: Clinical Trial Evaluating the Optimal Technique for Chest Tube Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F081016009
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2013-09

CONDITIONS: Chest Tube Removal
Keywords: Thoracotomy; Inspiration; Expiration; Chest Tube; pneumothorax; Method of chest tube removal
MeSH Terms: conditions — Respiratory Aspiration; Death; Pneumothorax | interventions — Exhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inspiration (Other)
  Interventions: Procedure: Chest tube pull on inspiration
- Expiration (Other)
  Interventions: Procedure: Expiration

INTERVENTIONS:
Procedure: Chest tube pull on inspiration — Pull chest tube on Inspiration
  Arms: Inspiration
Procedure: Expiration — Pull chest tube on Expiration
  Arms: Expiration

SUMMARY:
There are two commonly used methods to remove chest tubes following thoracotomy. One is to remove the chest tube at maximum inspiration, (patient is asked to take a deep breath in and hold it), and the other is to pull the chest tube at maximum expiration,(patient is asked to blow out as much air as they can can and hold it). There has been considerable discussion among Thoracic surgeons that one of these two methods may decrease the risk of pneumothorax, the most common complication associated with chest tube removal. The investigators will compare the two methods, and also identify risk factors of developing pneumothorax during chest tube removal.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are post thoracotomy, pulmonary resection (wedge, lobectomy, segmentectomy, pneumonectomy), AND
* Have at least one chest tube.

Exclusion Criteria:

* Less than 19 years old,
* With interstitial lung disease, OR
* Any patient intubated.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pneumothorax | Within 4 hours after chest tube removal

SECONDARY OUTCOMES:
Morbidity | 4 hours after chest tube removal

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Cerfolio, MD, Principal Investigator — University of Alabama at Birmingham, Department of Surgery
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States